CLINICAL TRIAL: NCT00392574
Title: A Multicenter, Double-Blind, Randomized Study to Compare The Safety and Efficacy of Prulifloxacin Versus Placebo in the Treatment of Acute Gastroenteritis in Adult Travelers
Brief Title: Safety and Efficacy of Prulifloxacin Versus Placebo in Traveler's Diarrhea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OPT-099-001
Record Dates: First submitted 2006-10-24; First posted 2006-10-26 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2010-08

CONDITIONS: Acute Gastroenteritis in Adult Travelers
Keywords: Gastroenteritis
MeSH Terms: conditions — Gastroenteritis | interventions — prulifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Prulifloxacin
  Interventions: Drug: Prulifloxacin
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prulifloxacin — Tablet
  Arms: 1
Drug: Placebo — Tablet
  Arms: 2

SUMMARY:
The objective of this pivotal Phase III study is to investigate the safety and efficacy of prulifloxacin versus placebo in the treatment of subjects with acute bacterial gastroenteritis.

DETAILED DESCRIPTION:
This double-blind trial will compare the safety and efficacy of prulifloxacin versus placebo in adult travelers with acute gastroenteritis characterized by diarrhea with one or more of the following signs or symptoms: nausea, vomiting, abdominal pain or cramping, fecal urgency, moderate to severe gas-related symptoms, or tenesmus of ≤72 hours duration.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Acute Bacterial Gastroenteritis;
* Traveler from Industrialized Country;
* Capable of giving Informed Consent

Exclusion Criteria:

* Fever (>100.3 degrees);
* Pregnant or Breast Feeding or Not using adequate birth control;
* Known or Suspected (co-)Infection with non-bacterial pathogen;
* Symptoms of Gastroenteritis of >72 hours;
* Bloody Diarrhea;
* Concomitant antibacterial with activity against enteric bacterial pathogens;
* History of IBD;
* Unable/Unwilling to comply with study protocol;
* > 2 doses of anti-diarrheal medication within 24 hours;
* Antimicrobial Treatment within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2006-08; Primary Completion 2008-02 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Time to last unformed stool | Study days 1-3

SECONDARY OUTCOMES:
Clinical cure based on relief of signs and symptoms | Study days 1-3
Microbiologic eradication rates | Study days 1-3

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Dupont, MD, Study Director — University of Texas
Locations (1):
- INC Research, New Hope, Pennsylvania, United States